CLINICAL TRIAL: NCT03938090
Title: Multimodality Assessment of Acute and Long Term Response to Optimised MultiSite Pacing Cardiac Resynchronisation (MSP CRT) Devices Compared to Biventricular (BiV) CRT, in Patients With Heart Failure
Brief Title: Optimised MultiSite Pacing Vector Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Severe delay in getting ethics/R&D approval, Covid delays in initiating study and enrolment. Lack of fellow support for continuing study. After 3-4 years delay, concepts now
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 012604
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Left Bundle-Branch Block; Systolic Dysfunction
Keywords: Cardiac Resynchronization Therapy; MultiSite Pacing
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, two-arm, randomized 1:1, crossover study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard biventricular pacing (Placebo Comparator): Cardiac resynchronization therapy (CRT) devices will be programmed as per standard biventricular pacing settings
  Interventions: Device: Standard biventricular pacing
- Optimised MultiSite Pacing (MSP) (Active Comparator): Cardiac resynchronization therapy (CRT) devices will be programmed as per optimal MSP programming settings; determined by greatest change in dP/dtmax and narrowest QRS duration.
  Interventions: Device: Optimised MultiSite Pacing

INTERVENTIONS:
Device: Optimised MultiSite Pacing — The intervention includes using optimal programming settings with MultiSite pacing configurations via the patient's CRT device. The device in use is the same for each arm, the only changes are the programming settings.
  Arms: Optimised MultiSite Pacing (MSP)
Device: Standard biventricular pacing — Conventional programming settings using biventricular pacing will be used
  Arms: Standard biventricular pacing

SUMMARY:
The objective of this clinical investigation is to evaluate the clinical benefits of an MultiSite pacing (MSP) with patient specific left ventricular vector optimization in patients receiving cardiac resynchronization therapy (CRT) after 6 months of therapy.

This clinical investigation is a single-center, prospective, two-arm, randomized 1:1, crossover study designed to evaluate the effectiveness of Optimized MSP CRT compared to conventional bi-ventricular pacing.

Data will be collected at enrolment, CRT implant procedure, hospital pre-discharge, one, three and six months post implant. Enrolment data collection will include demographics, cardiovascular history, medication, echocardiography measurements, heart failure quality of life questionnaire and six minute walk test distance.

CRT implant procedure data collection will include implanted system information, lead location and conduction times. The electrical conduction recording procedure will include surface ECG and device electrogram (EGM) recordings during various MSP vector pacing configurations at the time of CRT device implant.

Patients will also undergo simultaneous invasive pressure measurements using a left ventricular pressure wire to allow haemodynamic measurements (dP/dtmax) during various MSP vector pacing configurations.

Optimal MSP programming settings will be determined by the narrowest QRS duration recorded by 12 lead ECG and the greatest change in dP/dtmax by pressure wires study.

In a subgroup of patients (approximately 25 patients), non-invasive electrical activation data will be collected with electrocardiographic imaging (ECGi) within 45 days of the implant procedure.

Patients will then be randomized 1:1 to receive either standard biventricular pacing or Optimized MSP at their one-month follow-up (± 15 days) visit.

At the 3 months (± 15 days) post randomization follow up visit, data collection will include surface ECG, EGMs, echocardiographic parameters and quality of life questionnaire. The patients will then undergo cross-over to the alternate randomization group with programming adjusted accordingly.

At the final, 6 months (± 15 days) post randomization follow-up visit, data collection will include surface ECG, EGMs, echocardiographic parameters and quality of life questionnaire. This will mark the completion of the study for each patient.

The expected duration of enrolment is 18 months. The total duration of the clinical investigation is expected to be 25 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Heart Failure (NYHA class I-IV) with QRS duration of 150ms or more with left bundle branch block and LVEF of 35% or less despite optimal medical therapy.
* Patients above 18 years of age
* Able to provide informed consent and willing to comply with study requirements
* Intrinsic QRS duration ≥ 150 ms
* Sinus (or atrial paced) rhythm with intact AV conduction (PR interval ≤250 ms)

Exclusion Criteria:

* Resting heart rate > 100 bpm
* High degree AV Block (2nd or 3rd degree AV block)
* Documented persistent atrial arrhythmia at the moment of enrolment or patients not likely to remain in sinus (or atrial paced) rhythm for the duration of the study
* Patients scheduled for AV node ablation to treat atrial arrhythmias
* Recent (< 3 months) myocardial infarction, catheter ablation, electrolyte imbalance, or any condition within the last 90 days that would contraindicate CRT programming changes in the opinion of the investigator
* Women who are pregnant or plan to become pregnant during the study course
* Known left ventricular thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Echocardiographic clinical response | 3 and 6 months post randomization
  Response to optimised MSP CRT compared to BiV CRT defined by LV systolic volume reduction of greater than 15% (indicative of "reverse remodelling") at completion of follow up.

SECONDARY OUTCOMES:
Acute changes in surface ECG QRS duration and morphology | Acute change in QRS duration with pacing compared to intrinsic QRS duration, measured during pacing programming protcol at device implant
  QRS duration changes with CRT programming optimisation
Acute change in LV dP/dtmax | Acute change in LV dP/dtmax with pacing compared to intrinsic rhythm, measured during pacing programming protcol at device implant
  Changes in LV contractility as assessed by pressure wire
Change in exercise capacity by 6MWT distance | Pre-implant, 3 and 6 months post randomization
  6 minute walk test distance
Change in NYHA functional class | Pre-implant, 3 and 6 months post randomization
  New York Heart Association Functional class

OTHER OUTCOMES:
Sub-group outcome: assessment of LV activation timings with ECGi | 1 month post implant
  Electrocardiographic imaging

CONTACTS AND LOCATIONS:
Overall Officials: Anthony WC Chow, MBBS BSc MD, Principal Investigator — Study Chief Investigator
Locations (1):
- St Bartholomew's Hospital, Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared with other researchers